CLINICAL TRIAL: NCT05417269
Title: A Phase I/II Dose Escalation/Adaptive Design Study to Evaluate the Safety and Efficacy of IMCY-0141 in Patients With Relapsing Remitting-Multiple Sclerosis (RR-MS)
Brief Title: IMCY-0141 Safety and Efficacy in Multiple Sclerosis - ISEMIS Study
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imcyse SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMCY-MS-001; 2021-004974-67 (EudraCT Number)
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: RR-MS; Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis; Synthetic peptide
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Intervention Model Description: The study will be conducted under a Bayesian adaptive design approach comprising of two phases:
  * Phase I where 3 IMCY-0141 doses will be administered following a dose escalation approach. An IDMC safety assessment will allow the escalation from lower to upper dose.
  * Phase IIa leading to a preliminary estimate of the efficacy of each dose and determination of promising doses. The 2 doses that emerge as most promising will be recommended to advance to Phase IIb, where final efficacy will be judged, again relative to placebo. The least promising dose may be dropped, at the discretion of the trial's IDMC.
  All told, Phase II will enrol patients who will be randomized to IMCY-0141 or placebo or DMF. At the conclusion of Phase IIb, determined doses will be labelled effective.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a two-step study with a phase I, open-label, dose escalation clinical trial to evaluate the safety of three IMCY-0141 doses followed by a phase II, double-blind, randomized study with an adaptive design to determine if any IMCY-0141 doses offer superior efficacy relative to placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 - Phase I (IMCY-0141 Dose 1) (Experimental): The first dose (Cohort 1) will consist of the administration of 150 μg of peptide (IMCY-0141) in two separate injections of 75 μg each (500μl each).
  Interventions: Drug: IMCY-0141
- Cohort 2 - Phase I (IMCY-0141 Dose 2) (Experimental): The second dose (Cohort 2) will consist of the administration of 450 μg of peptide (IMCY-0141) in two separate injections of 225 μg each (500μl each).
  Interventions: Drug: IMCY-0141
- Cohort 3 - Phase I (IMCY-0141 Dose 3) (Experimental): The third dose (Cohort 3) will consist of the administration of 1350 μg of peptide (IMCY-0141) in two separate injections of 675 μg each (500μL each).
  Interventions: Drug: IMCY-0141
- Group 1 - Phase II (IMCY-0141 Dose 1) (Experimental): Administration of IMCY-0141, 150 μg combined with alum adjuvant.
  Interventions: Drug: IMCY-0141
- Group 2 - Phase II (IMCY-0141 Dose 2) (Experimental): Administration of IMCY-0141, 450 μg combined with alum adjuvant.
  Interventions: Drug: IMCY-0141
- Group 3 - Phase II (IMCY-0141 Dose 3) (Experimental): Administration of IMCY-0141, 1350 μg combined with alum adjuvant.
  Interventions: Drug: IMCY-0141
- Group 4 (Placebo Group) - Phase II (Placebo Comparator): Administration of placebo combined with alum adjuvant.
  Interventions: Drug: Placebo
- Group 5 (Active Control Group) - Phase II (Active Comparator): Parallel, Open-Label, Active Control Group Oral administration of Dimethyl Fumarate (DMF) given according to its SmPC for the whole duration of the study.
  Interventions: Drug: Dimethyl Fumarate

INTERVENTIONS:
Drug: IMCY-0141 — The investigational medicinal product (IMP) consists in a small synthetic peptide (23 amino acids - IMCY-0141) combining a known human epitope of MOG flanked with a thioredox motif, presented in the form of a freeze-dried sterile powder and diluent for subcutaneous (SC) administration. The diluent includes the adjuvant aluminium hydroxide (alum) at a concentration of 900 μg/mL. Treatment will be injected within 4h of resuspension of the powder with the diluent.
  Treatment will consist of 6 immunizations (separated by 14 days) of the IMP by SC injection in the upper arm, in the region of the triceps (lateral part of the arm, midway between the elbow and the shoulder). Half of the dose to be administered will be injected concomitantly in both arms.
  Other Names: Imotope
  Arms: Cohort 1 - Phase I (IMCY-0141 Dose 1); Cohort 2 - Phase I (IMCY-0141 Dose 2); Cohort 3 - Phase I (IMCY-0141 Dose 3); Group 1 - Phase II (IMCY-0141 Dose 1); Group 2 - Phase II (IMCY-0141 Dose 2); Group 3 - Phase II (IMCY-0141 Dose 3)
Drug: Placebo — The placebo will be administered by subcutaneous route, once every two weeks for 6 times. Placebo will be administered to patients randomized in the "placebo" group during Phase II only.
  Arms: Group 4 (Placebo Group) - Phase II
Drug: Dimethyl Fumarate — Dimethyl Fumarate (DMF) will be given orally, according to its SmPC for the whole duration of the study.
  Dimethyl Fumarate (DMF) will be administered to patients randomized in the active control group during Phase II only.
  Other Names: DMF
  Arms: Group 5 (Active Control Group) - Phase II

SUMMARY:
The IMCY-MS-001 study is a study to test a new experimental drug, IMCY-0141, for the treatment of Relapsing-Remitting Multiple Sclerosis (RR-MS).

The pathophysiology of MS with known myelin autoantigens and T cell epitopes makes this disease a particularly attractive indication for development of an immunotherapeutic based on the Imcyse technology.

Based on the unique mechanism of action of the drug, IMCY-0141 administered as early as possible after confirmation of the diagnosis may potentially switch-off the autoimmune process and limit the corresponding myelin destruction. Newly (recently) diagnosed patients will be targeted to tackle the disease at its onset.

Before launching any efficacy studies, safety of IMCY-0141 in MS patients must be evaluated with a phase I, open-label, dose escalation clinical trial to evaluate the safety of three IMCY-0141 doses followed by a phase II, double-blind, randomized study with an adaptive design to determine if any IMCY-0141 dose(s) offer superior efficacy relative to placebo and to assess immune responses and biomarker data as potential early predictors of efficacy of IMCY-0141 in adults presenting with RR-MS.

DETAILED DESCRIPTION:
The Sample Size determined for this study is as follows:

Phase I:

A total of 12 patients (4 patients in each of 3 dose cohorts) are planned to be enrolled. The study sample size has been estimated as adequate to provide a reliable safety assessment of the tested doses. All primary, secondary and exploratory endpoints will be summarized by descriptive statistics (continuous variables) or frequency tables (categorical variables), by dose group and overall. Additional patients may be enrolled if requested by the IDMC (Independent Data Monitoring Committee).

Phase II:

The sample size estimation is based on the total cumulative number of CUAL observed on brain MRI scans from week 12 till week 36. The study sample size has been estimated as adequate to determine if any IMCY-0141 doses offer superior efficacy (as measured by CUAL) relative to placebo. Using the negative binomial model for CUAL, a maximum total of 150 patients are planned to be enrolled (including the 12 patients enrolled in phase I), with 30 patients randomized to each of five groups:

* Placebo
* IMCY-0141 dose 1
* IMCY-0141 dose 2
* IMCY-0141 dose 3
* DMF (open label)

During the adaptive design phase (Phase IIa), a minimum of 40 patients will be enrolled (with 8 patients randomized to each of five groups) and analyzed along with the 12 phase I patients as detailed here:

* Placebo: 8 patients
* IMCY-0141 dose 1: 8 patients + 4 phase I patients
* IMCY-0141 dose 2: 8 patients + 4 phase I patients
* IMCY-0141 dose 3: 8 patients + 4 phase I patients
* DMF (open label) : 8 patients

During the Phase IIb part, up to 98 additional patients will be enrolled in order to get up to 150 patients spread over the groups selected for Phase IIb, with a maximum 30 patients randomized to DMF. These sample sizes are sufficient to deliver Type I errors less than 5% in our chosen null scenarios, and unconditional powers greater than 75% and conditional powers greater than 90% in our two alternative scenarios.

ELIGIBILITY:
Inclusion Criteria (Phase I and II):

1. Male or female between 18 and and 45 years old.
2. RR-MS according to the 2017 revisions of the McDonald Criteria.
3. Patients should be newly diagnosed or have a disease duration ≤ 3 years.
4. If not newly diagnosed, patients should have at least one documented clinical relapse in the last 12 months.
5. Patients should present with at least 1 Gadolinium-enhancing (Gd+) T1-weighted lesion OR at least 2 new or enlarging T2-weighted lesions at screening MRI compared to a reference scan in the last 6 months.
6. No background MS treatment at the time of study treatment start (refer to exclusion criteria for details about authorized washout period for some first line treatment).
7. EDSS ≤ 5.0 at screening.
8. Women of childbearing potential (1) should use an highly effective contraception method (2) from screening and for the whole duration of the study. (1) Of child-bearing potential is defined as being post onset of menarche and not meeting any of the following conditions:

   * Menopausal for at least 2 years (follicle-stimulating hormone within menopausal range),
   * Having undergone bilateral tubal ligation at least 1 year previously
   * Having undergone bilateral oophorectomy or hysterectomy. (2) HIGHLY EFFECTIVE contraceptive measures acceptable for the whole duration of the study have been defined based on the CTFGs recommendations on contraception and are the following:
   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal),
   * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).
   * Intrauterine device (IUD)
   * intrauterine hormone-releasing system (IUS)
   * Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least 6 months prior to the patient's entry into the study
   * Abstinence or absence of sexual relations with men.
9. Ability to understand and comply with research requirements and procedures, in opinion of investigator (Signed Informed Consent)

Exclusion Criteria (Phase I and II):

1. Secondary or primary progressive multiple sclerosis and late onset multiple sclerosis (LOMS).
2. Findings on brain MRI scan indicating any clinically significant brain abnormality like:

   * Doubts about MS diagnosis (based on clinically or imaging abnormalities)
   * PML cases (positive PML checklist according to "suspected PML case adjudication instructions")
   * Co-morbidities influencing the MS disease evolution (i.e. Tumor, large infarction, CSF obstruction)
3. Patient has complete transverse myelitis or bilateral optic neuritis.
4. Systemic corticosteroids or adrenocorticotropic hormone (ACTH) without chronic use within 30 days prior to screening MRI.
5. Treatment with rituximab, ocrelizumab, mitoxantrone, or lymphocyte depleting therapies (e.g., alemtuzumab, anti-CD4, cladribine, cyclophosphamide, total body irradiation, bone marrow transplantation) within 48 weeks prior to study treatment start.
6. Use of lymphocyte trafficking blockers (e.g., natalizumab, fingolimod) within 24 weeks prior to study treatment start.
7. Treatment with β-interferons or glatiramer acetate within 4 weeks prior to study treatment start.
8. Treatment with teriflunomide within 12 weeks prior to study treatment start.
9. Exposure to dimethyl fumarate within 6 months prior to study treatment start.
10. Any investigational drug within the past 6 months at the time of study treatment start.
11. Immunosuppressive therapy including chronic use of systemic steroids in past year. Topical, inhalational or intranasal corticosteroids are allowed.
12. Primary or secondary immune deficiency disorders with the exception of well-controlled diabetes or thyroid disorder.
13. Patients with combined other auto-immune or inflammatory disorders.
14. Have signs or symptoms of active or long COVID infection or a positive COVID PCR test during the screening period. In the case of PCR positivity, a reswabbing will be done. If reswabbing returns a negative result, the initiation of study treatment can occur.
15. Have evidence of current or past human immunodeficiency virus (HIV-1 and 2), Hepatitis B or Hepatitis C infection: HBsAg+ or anti-HBc+; anti-HCV+ (unless the polymerase chain reaction [PCR] for HBV DNA (hepatitis B) or HCV RNA (hepatitis C) is negative according to local procedure).
16. Current signs or symptoms of infection at time of study treatment start or within 2 weeks prior to planned administration of the study product or intravenous antibiotics within 2 months prior to the first planned administration of the study product.
17. Live, attenuated vaccine within 3 months prior to the first planned administration of the study product.
18. Inability to comply with MRI scanning, including contraindications to MRI such as known allergy to gadolinium contrast media, claustrophobia, presence of a pacemaker, cochlear implants, ferromagnetic devices or clips, intracranial vascular clips, insulin pumps, nerve stimulators.
19. Any other significant disease, disorder or finding which may significantly increase the risk to the patient because of participation in the study, affect the ability of the patient to participate in the study or impair interpretation of the study data.
20. Patients with a known hypersensitivity to any component of the drug product.
21. Patients with psychiatric or cognitive disorders.
22. History of MS related seizures not adequately controlled by medications.
23. History of cancer, except adequately treated basal cell or squamous cell carcinoma of the skin (no more than 3 lesions requiring treatment in lifetime) or carcinoma in situ/cervical intraepithelial neoplasia of the uterine cervix, unless considered cured > 5 years
24. Abnormal renal function defined by creatinine clearance ≤ 60 ml/min/1.73m2.
25. Patient with total lymphocytes count < 1000/mm3.
26. Patient with abnormal hepatic function defined as any liver enzyme > 3 ULN, bilirubin > 3 ULN with exception of Gilbert Syndrome.
27. Breastfeeding/lactating or pregnant women.

Exclusion Criteria specific for Phase I:

1. Patient HLA DRB1*03:01 positive

Exclusion Criteria specific for Phase II:

1. Patients already included in Phase I

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ph I Primary safety endpoint (1) - Solicited injection site and systemic AEs | Up to 36 weeks
  Occurrence, intensity and relationship of any solicited injection site and systemic adverse events (AEs) during a 7-day follow-up period (i.e., day of study product administration and 6 subsequent days) after each IMCY-0141 administration analysing local injection site and systemic adverse events, clinical and laboratory data.
Ph I Primary safety endpoint (2) - Unsolicited injection site and systemic AEs | Up to 36 weeks
  Occurrence, intensity and relationship of any unsolicited injection site (local) and systemic AEs occurring throughout the study period.
Ph I Primary safety endpoint (3) - All SAEs | Up to 36 weeks
  Occurrence and relationship of all serious adverse events (SAEs) occurring throughout the study period.
Ph I Primary safety endpoint (4) - Abnormalities on different parameters | Up to 36 weeks
  Occurrence and relationship of any abnormality in physical examination, vital signs, 12-lead ECG, MRI, haematological and biochemical laboratory parameters.
Ph II Primary efficacy endpoint - Number of CUAL | Week 12 to Week 36
  Total cumulative number of CUAL observed on brain MRI scans (centralized reading) from week 12 till week 36 vs placebo.

SECONDARY OUTCOMES:
Ph I/II Secondary endpoint (1) - Relapse rate | At Week 36
  Annualized relapse rate at week 36 vs baseline
Ph I/II Secondary endpoint (2) - Relapse-free rate | At Week 36
  Proportion of relapse-free patients at week 36 vs baseline
Ph I/II Secondary endpoint (3) - EDSS Score | At Week 36
  EDSS score at week 36 vs screening
Ph I/II Secondary endpoint (4) - Neurofilament light chains levels | Up to 36 weeks
  Neurofilament light chains levels in the serum of the patient (sNfL) at baseline, weeks 2, 4, 6, 8, 10, 12, 24 and 36.
Ph II Secondary endpoint (1) - Solicited injection site and systemic AEs | Up to 36 weeks
  Occurrence, intensity and relationship of any solicited local and systemic adverse event (AE) during a 7-day follow-up period (i.e., day of study drug administration and 6 subsequent days) after each IMCY-0141 administration.
Ph II Secondary endpoint (2) - Unsolicited injection site and systemic AEs | Up to 36 weeks
  Occurrence, intensity and relationship of any unsolicited injection site (local) and systemic AEs occurring throughout the study period.
Ph II Secondary endpoint (3) - All SAEs | Up to 36 weeks
  Occurrence and relationship of all serious adverse events (SAEs) occurring throughout the study period.
Ph II Secondary endpoint (4) - Abnormalities on different parameters | Up to 36 weeks
  Occurrence, intensity and relationship of any abnormality in physical examination, vital signs, 12-lead ECG, MRI, haematological and biochemical laboratory parameters.

OTHER OUTCOMES:
To assess the disease activity and the efficacy of IMCY-0141 on MRI parameters and if any IMCY-0141 dose(s) offer superior efficacy. | Up to 36 weeks
  Measured by cumulative number of CUAL, number of new Gadolinium-enhancing T1 lesions, number of active (new or enlarging) T2/FLAIR lesions, number of persistent Gadolinium enhancing T1 lesions vs baseline and number of shrinking FLAIR lesions versus baseline.
To assess the disease activity | Up to 36 weeks
  Measured by volume change versus baseline in T2/FLAIR lesions, Gadolinium-enhancing T1 lesions, shrinking FLAIR lesions and Brain (White matter, grey matter, cortical grey matter, lateral, thalamus)
To evaluate and characterize the MOG-specific CD4+ T cells induced by IMCY-0141 and its impact on autoreactive T-cell responses specific for myelin proteins. | Up to 36 weeks
  Changes in cytolytic CD4+ T cell response specific for IMCY-0141, in CD4+ and CD8+ effector T cell responses specific for myelin proteins MOG and/or PLP
Impact of IMCY-0141 on auto-antibodies against myelin proteins (MOG,PLP) | Up to 36 weeks
  Detection of change in MS associated auto-antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Vitalie LISNIC, Prof., Principal Investigator — ARENSIA Exploratory Medicine, Moldova
Locations (1):
- Republican Clinical Hospital, ARENSIA Exploratory Medicine, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malek Abrahimians E, Carlier VA, Vander Elst L, Saint-Remy JM. MHC Class II-Restricted Epitopes Containing an Oxidoreductase Activity Prompt CD4(+) T Cells with Apoptosis-Inducing Properties. Front Immunol. 2015 Sep 2;6:449. doi: 10.3389/fimmu.2015.00449. eCollection 2015. PMID 26388872
- [Background] Carlin BP, Louis TA. Bayesian Methods for Data Analysis, 3rd ed. 2009; Boca Raton, FL: CRC Press.
- [Background] Cohen JA, Coles AJ, Arnold DL, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Fisher E, Brinar VV, Giovannoni G, Stojanovic M, Ertik BI, Lake SL, Margolin DH, Panzara MA, Compston DA; CARE-MS I investigators. Alemtuzumab versus interferon beta 1a as first-line treatment for patients with relapsing-remitting multiple sclerosis: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1819-28. doi: 10.1016/S0140-6736(12)61769-3. Epub 2012 Nov 1. PMID 23122652
- [Background] Coles AJ, Twyman CL, Arnold DL, Cohen JA, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Miller T, Fisher E, Sandbrink R, Lake SL, Margolin DH, Oyuela P, Panzara MA, Compston DA; CARE-MS II investigators. Alemtuzumab for patients with relapsing multiple sclerosis after disease-modifying therapy: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1829-39. doi: 10.1016/S0140-6736(12)61768-1. Epub 2012 Nov 1. PMID 23122650
- [Background] Committee for Medicinal Products for Human Use (CHMP) of the European Medicines Agency. Guideline on the clinical investigation of medicinal products for the treatment of multiple sclerosis. CHMP/771815/2011 Rev. 2. Effective date 1 October 2015.
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Friese MA, Fugger L. Autoreactive CD8+ T cells in multiple sclerosis: a new target for therapy? Brain. 2005 Aug;128(Pt 8):1747-63. doi: 10.1093/brain/awh578. Epub 2005 Jun 23. PMID 15975943
- [Background] Goldenberg MM. Multiple sclerosis review. P T. 2012 Mar;37(3):175-84. No abstract available. PMID 22605909
- [Background] Guo X, Carlin BP. Separate and joint modeling of longitudinal and event time data using standard computer packages. The American Statistician; 2004; 58, 16-24.
- [Background] Johnson KP, Brooks BR, Cohen JA, Ford CC, Goldstein J, Lisak RP, Myers LW, Panitch HS, Rose JW, Schiffer RB. Copolymer 1 reduces relapse rate and improves disability in relapsing-remitting multiple sclerosis: results of a phase III multicenter, double-blind placebo-controlled trial. The Copolymer 1 Multiple Sclerosis Study Group. Neurology. 1995 Jul;45(7):1268-76. doi: 10.1212/wnl.45.7.1268. PMID 7617181
- [Background] Kampman MT, Brustad M. Vitamin D: a candidate for the environmental effect in multiple sclerosis - observations from Norway. Neuroepidemiology. 2008;30(3):140-6. doi: 10.1159/000122330. Epub 2008 Apr 2. PMID 18382112
- [Background] Kappos L, Antel J, Comi G, Montalban X, O'Connor P, Polman CH, Haas T, Korn AA, Karlsson G, Radue EW; FTY720 D2201 Study Group. Oral fingolimod (FTY720) for relapsing multiple sclerosis. N Engl J Med. 2006 Sep 14;355(11):1124-40. doi: 10.1056/NEJMoa052643. PMID 16971719
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] McCarthy DP, Richards MH, Miller SD. Mouse models of multiple sclerosis: experimental autoimmune encephalomyelitis and Theiler's virus-induced demyelinating disease. Methods Mol Biol. 2012;900:381-401. doi: 10.1007/978-1-60761-720-4_19. PMID 22933080
- [Background] McKay KA, Kwan V, Duggan T, Tremlett H. Risk factors associated with the onset of relapsing-remitting and primary progressive multiple sclerosis: a systematic review. Biomed Res Int. 2015;2015:817238. doi: 10.1155/2015/817238. Epub 2015 Jan 31. PMID 25802867
- [Background] National Cancer Institute (NCI); U.S. Department of health and human services, National Institutes of Health. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Published: May 28, 2009 (v4.03: June 14, 2010).
- [Background] National Multiple Sclerosis Society. Who Gets MS?. http://www.nationalmssociety.org/aboutmultiple-sclerosis/what-we-know-about-ms/who-gets-ms/index.aspx. Accessed 30 March 2016.
- [Background] Noonan CW, Williamson DM, Henry JP, Indian R, Lynch SG, Neuberger JS, Schiffer R, Trottier J, Wagner L, Marrie RA. The prevalence of multiple sclerosis in 3 US communities. Prev Chronic Dis. 2010 Jan;7(1):A12. Epub 2009 Dec 15. PMID 20040227
- [Background] Olsson T, Boster A, Fernandez O, Freedman MS, Pozzilli C, Bach D, Berkani O, Mueller MS, Sidorenko T, Radue EW, Melanson M. Oral ponesimod in relapsing-remitting multiple sclerosis: a randomised phase II trial. J Neurol Neurosurg Psychiatry. 2014 Nov;85(11):1198-208. doi: 10.1136/jnnp-2013-307282. Epub 2014 Mar 21. PMID 24659797
- [Background] Polman CH, O'Connor PW, Havrdova E, Hutchinson M, Kappos L, Miller DH, Phillips JT, Lublin FD, Giovannoni G, Wajgt A, Toal M, Lynn F, Panzara MA, Sandrock AW; AFFIRM Investigators. A randomized, placebo-controlled trial of natalizumab for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):899-910. doi: 10.1056/NEJMoa044397. PMID 16510744
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Randomised double-blind placebo-controlled study of interferon beta-1a in relapsing/remitting multiple sclerosis. PRISMS (Prevention of Relapses and Disability by Interferon beta-1a Subcutaneously in Multiple Sclerosis) Study Group. Lancet. 1998 Nov 7;352(9139):1498-504. PMID 9820297
- [Background] Rosati G. The prevalence of multiple sclerosis in the world: an update. Neurol Sci. 2001 Apr;22(2):117-39. doi: 10.1007/s100720170011. PMID 11603614
- [Background] Rudick RA, Panzara MA. Natalizumab for the treatment of relapsing multiple sclerosis. Biologics. 2008 Jun;2(2):189-99. doi: 10.2147/btt.s1956. PMID 19707353
- [Background] Selmaj K, Li DK, Hartung HP, Hemmer B, Kappos L, Freedman MS, Stuve O, Rieckmann P, Montalban X, Ziemssen T, Auberson LZ, Pohlmann H, Mercier F, Dahlke F, Wallstrom E. Siponimod for patients with relapsing-remitting multiple sclerosis (BOLD): an adaptive, dose-ranging, randomised, phase 2 study. Lancet Neurol. 2013 Aug;12(8):756-67. doi: 10.1016/S1474-4422(13)70102-9. Epub 2013 Jun 11. PMID 23764350
- [Background] Sormani MP, Miller DH, Comi G, Barkhof F, Rovaris M, Bruzzi P, Filippi M. Clinical trials of multiple sclerosis monitored with enhanced MRI: new sample size calculations based on large data sets. J Neurol Neurosurg Psychiatry. 2001 Apr;70(4):494-9. doi: 10.1136/jnnp.70.4.494. PMID 11254773
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Varhaug KN, Barro C, Bjornevik K, Myhr KM, Torkildsen O, Wergeland S, Bindoff LA, Kuhle J, Vedeler C. Neurofilament light chain predicts disease activity in relapsing-remitting MS. Neurol Neuroimmunol Neuroinflamm. 2017 Nov 28;5(1):e422. doi: 10.1212/NXI.0000000000000422. eCollection 2018 Jan. PMID 29209636
- [Background] Varhaug KN, Torkildsen O, Myhr KM, Vedeler CA. Neurofilament Light Chain as a Biomarker in Multiple Sclerosis. Front Neurol. 2019 Apr 5;10:338. doi: 10.3389/fneur.2019.00338. eCollection 2019. PMID 31024432
- [Background] Weiner HL. Multiple sclerosis is an inflammatory T-cell-mediated autoimmune disease. Arch Neurol. 2004 Oct;61(10):1613-5. doi: 10.1001/archneur.61.10.1613. No abstract available. PMID 15477521
- [Background] Zhu H, Lakkis H. Sample size calculation for comparing two negative binomial rates. Stat Med. 2014 Feb 10;33(3):376-87. doi: 10.1002/sim.5947. Epub 2013 Aug 23. PMID 24038204